CLINICAL TRIAL: NCT03307837
Title: A Phase 1/Single Ascending Dose (SAD) Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of a Single Intraoperative Administration of CA-008 in Subjects Undergoing Correction of Hallux Valgus Deformity
Brief Title: A Phase 1 Study of Intraoperative Administration of CA-008 for the Correction of Hallux Valgus Deformity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concentric Analgesics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CA-PS-2017-101
Record Dates: First submitted 2017-10-03; First posted 2017-10-12 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Hallux Valgus Deformity
Keywords: Unilateral Transpositional First Metatarsal Osteotomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- CA-008 Cohort 1 0.5 mg (Active Comparator): Intra-operative, local administration
  Interventions: Drug: CA-008
- CA-008 Cohort 2 1 mg (Active Comparator): Intra-operative, local administration
  Interventions: Drug: CA-008
- CA-008 Cohort 3 2 mg (Active Comparator): Intra-operative, local administration
  Interventions: Drug: CA-008
- CA-008 Cohort 4 3 mg (Active Comparator): Intra-operative, local administration
  Interventions: Drug: CA-008
- CA-008 Cohort 5 4.2 mg (Active Comparator): Intra-operative, local administration
  Interventions: Drug: CA-008
- Placebo (Placebo Comparator): Intra-operative, local administration of saline (equivalent volume in active comparator arm)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CA-008 — Local administration during surgery
  Arms: CA-008 Cohort 1 0.5 mg; CA-008 Cohort 2 1 mg; CA-008 Cohort 3 2 mg; CA-008 Cohort 4 3 mg; CA-008 Cohort 5 4.2 mg
Drug: Placebo — Local administration during surgery
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, single ascending dose, sequential-group Phase 1 study. The study will be conducted utilizing a cohort design, with sequential groups of 8 subjects. Within each dose cohort, 6 subjects will be randomized to active, and 2 will be randomized to placebo.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled, single ascending dose, sequential-group Phase 1 study.

The study will be conducted utilizing a cohort design, with sequential groups of 8 subjects. Within each dose cohort, 6 subjects will be randomized to active, and 2 will be randomized to placebo. Placebo patients from each cohort were pooled for analysis. The initial cohort will receive the lowest planned dose of CA-008, and sequential cohorts will receive escalating doses of CA-008 in a fixed volume of administration. There will be at least a 6-day period between cohorts, in order to ensure a minimum of 3 days to review safety data from the last subject in a cohort and to allow the meeting of the Data Monitoring Committee (DMC) to review the safety data from the entire cohort prior to a making decision for dose escalation. Dose escalation rules will be protocol defined.

Subjects will be undergoing unilateral transpositional first metatarsal osteotomy for the correction of hallux valgus deformity (bunionectomy). In accordance with standard of care, subjects will receive regional anesthesia (MAYO block) with 0.5% bupivacaine. Prior to wound closure, 10 mL of study drug will be injected into the soft tissues and periosteum of the surgical site.

After the surgery, subjects will be monitored for 48 hours at the trial site. Safety and efficacy evaluations will be performed as described herein. Subjects will be required to meet certain pre-specified criteria prior to discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 - 65 years old, inclusive.
2. Planning to undergo a primary unilateral first metatarsal bunionectomy repair, without collateral procedures.
3. Be American Society of Anesthesiology (ASA) physical Class 1 or 2.
4. In good health and capable of undergoing a bunionectomy under regional anesthesia.
5. No additional planned surgeries other than a bunionectomy during the course of the study.
6. Male subjects must be either sterile (surgically or biologically), or commit to an acceptable method of birth control while participating in the study.
7. Female subjects are eligible only if all of the following apply:

   1. Not pregnant (female subject of child bearing potential must have a negative serum pregnancy tests at screening and negative urine pregnancy test before surgery);
   2. Not lactating;
   3. Not planning to become pregnant during the study;
   4. Be surgically sterile; or at least two years post-menopausal; or have a monogamous partner who is surgically sterile; or is practicing double-barrier contraception; or practicing abstinence (must agree to use double-barrier contraception in the event of sexual activity); or using an insertable, injectable, transdermal, or combination oral contraceptive approved by the FDA for greater than 2 months prior to screening visits and commits to the use of an acceptable form of birth control for the duration of the study and for 30 days from completion of the study.
8. Have a body mass index ≤ 35 kg/m2.
9. Willing and able to sign the informed consent form (ICF) approved by the Institutional Review Board (IRB).
10. Willing and able to complete the study procedures and pain scales, and to communicate meaningfully in English with study personnel.

Exclusion Criteria:

1. Subjects with a history of hypertension, cardiovascular disease and a history of cerebrovascular events.
2. Subjects with concurrent painful conditions that may require analgesic treatment during the study period, or, in the opinion of the Investigator, may confound post-operative pain assessments.
3. Have been receiving or have received chronic opioid therapy defined as greater than 15 morphine equivalents units per day for greater than 3 out of 7 days per week over a one-month period within 12 months of study treatment initiation.
4. Have a known allergy or intolerance to the following medications or related substances: capsaicin, chili peppers, propofol, bupivacaine, benzodiazepines, midazolam, oxycodone, or ondansetron.
5. Have a clinically significant abnormal clinical laboratory test value according to the judgment of the investigator.
6. Have, as determined by the investigator or the study's medical monitor, a history or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, or other condition that would preclude participation in the study.
7. Use concurrent therapy that could interfere with the evaluation of efficacy or safety, such as any drugs which, in the investigator's opinion, may exert significant analgesic properties or act synergistically with CA-008.
8. Use of disallowed pain medications within 2 days prior to Day 1 (NSAIDs, COX-2 inhibitors, tramadol, ketamine, clonidine, gabapentin, pregabalin, or cannabinoids).
9. Use of central nervous system (CNS) active drugs such as benzodiazepines, tricyclic antidepressants, SNRIs, or SSRIs for pain within seven days prior to Day 1. These drugs are permitted for non-pain indications if the dose has been stable for at least 30 days prior to Day 1 and is planned to remain stable throughout the study. The use of lorazepam and other sleep medications, except those containing analgesic properties, is permitted.
10. Have evidence of a clinically significant 12-lead ECG abnormality according to the judgment of the investigator, including QTcF >450 for men and >470 for women.
11. Use of dietary supplements or over-the-counter (OTC) medications containing significant amounts of capsaicin within 1 day prior to Day 1, and throughout the hospitalization period.
12. Subjects with active cutaneous disease, or other disease, at the anticipated site of surgery.
13. History of peripheral vascular disease, sickle cell disease, vascular grafts, or vasospastic disorders.
14. Use of parenteral or oral corticosteroid(s) within 14 days prior to Day 1.
15. Known bleeding disorder or is taking agents affecting coagulation preoperatively. Deep venous thrombosis (DVT) prophylaxis of the surgeon's choice is permitted postoperatively.
16. A medical condition that in the investigator's opinion could adversely impact the subject's participation or safety, conduct of the study, or interfere with the pain assessments.
17. Diabetes mellitus.
18. Use of antihypertensive agent or diabetic regimen at a dose that has not been stable for at least 30 days, or which is not expected to remain stable throughout the study.
19. Use of digoxin, warfarin (see exception below), lithium, theophylline preparations, aminoglycosides, and all antiarrhythmics except beta-blockers, and use of anticonvulsants except benzodiazepines within 7 days prior to Day 1 and throughout the study. (Use of warfarin is allowed, at the investigator's discretion, for DVT prophylaxis after the surgery).
20. History of illicit drug use, or prescription medicine or alcohol abuse (regularly drinks > 4 units of alcohol per day; 8 oz. beer, 3 oz. wine, 1 oz. spirits) within the past 2 years, in the opinion of the Investigator.
21. Have positive results on the alcohol breath test indicative of alcohol abuse or urine drug screen indicative of illicit drug use (unless results can be explained by a current prescription or acceptable over-the-counter medication at screening as determined by the investigator) at screening, and/or prior to surgery.
22. Stable medication regimen for at least 14 days prior to the scheduled bunionectomy procedure, within 5 half-lives of the specific prior medication (or, if half-life is not known, within 48 hours) before dosing with study medication.
23. Participated in another clinical trial or used an investigational product within 30 days or five half-lives (whichever is longer) prior to the planned bunionectomy surgery, or is scheduled to receive an investigational product other than CA-008 while participating in the study.
24. Previously participated in a clinical study with CA-008 or capsaicin.
25. Subjects with peripheral neuropathies which would potentially confound the planned neurosensory testing.
26. Any past or current medical condition that in opinion of investigator, puts subject at undue safety risk for surgical complications or for use of the investigational product.
27. Subjects who donated blood or plasma within the 30 days prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Donovan, MD, Study Director — Concentric Analgesics
Locations (1):
- Lotus Clinical Research, LLC, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 40 enrolled participants, all 40 met inclusion criteria and were randomized to treatment.
Groups:
- CA-008 Cohort 1 0.5 mg; CA-008 Cohort 2 1 mg; CA-008 Cohort 3 2 mg; CA-008 Cohort 4 3 mg; CA-008 Cohort 5 4.2 mg: Active (CA-008) to Placebo
- Placebo: Placebo
Period: Overall Study
Arm/Group | CA-008 Cohort 1 0.5 mg | CA-008 Cohort 2 1 mg | CA-008 Cohort 3 2 mg | CA-008 Cohort 4 3 mg | CA-008 Cohort 5 4.2 mg | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 10
Completed | 5 | 5 | 5 | 6 | 6 | 8
Not Completed | 1 | 1 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- CA-008 Cohort 1 0.5 mg; CA-008 Cohort 2 1 mg; CA-008 Cohort 3 2 mg; CA-008 Cohort 4 3 mg; CA-008 Cohort 5 4.2 mg: CA-008: The active moiety of CA-008, capsaicin that has certain properties for treatment of post-operative pain.
- CA-008 Placebo: CA-008 Placebo: Placebo product
- Total: Total of all reporting groups
Arm/Group | CA-008 Cohort 1 0.5 mg | CA-008 Cohort 2 1 mg | CA-008 Cohort 3 2 mg | CA-008 Cohort 4 3 mg | CA-008 Cohort 5 4.2 mg | CA-008 Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (12.94) | 32.0 (6.78) | 40.3 (12.52) | 39.5 (12.94) | 34.3 (10.25) | 34.9 (7.82) | 35.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 6 | 6 | 5 | 8 | 34
  Male | 1 | 2 | 0 | 0 | 1 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 1 | 2 | 1 | 2 | 14
  Not Hispanic or Latino | 1 | 3 | 5 | 4 | 5 | 8 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 3 | 1 | 5 | 15
  White | 5 | 3 | 4 | 3 | 4 | 3 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Surgical Site Assessment
Description: Assessment of skin reactions to determine if any change from 24 to 48 hours.
Time Frame: 24 and 48 hours post infiltration
Population: Safety Population
Measure: Number; unit: Number of skin reactions
Groups:
- Cohort 1: CA-008 in 0.5 mg dose
- Cohort 2: CA-008 in 1 mg dose
- Cohort 3: CA-008 in 2 mg dose
- Cohort 4: CA-008 in 3 mg dose
- Cohort 5: CA-008 in 4.2 mg dose
- Placebo: Placebo administration
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Number of skin reactions | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Neurosensory Assessment
Description: Change in neurosensory assessments of the skin surrounding the incision.
Time Frame: 48 hours post infiltration
Population: Safety population
Measure: Number; unit: Number of neurosensory abnormalities
Groups:
- Cohort 1: CA-008 in doses of 0.5 mg
- Cohort 2: CA-008 in doses of 1 mg
- Cohort 3: CA-008 in doses of 2 mg
- Cohort 4: CA-008 in doses of 3 mg
- Cohort 5: CA-008 in doses of 4.2 mg
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Number of neurosensory abnormalities | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: 11-point (0-10) Numerical Pain Rating Scale (NPRS)
Description: Pain as assessed by a standard 11-point (0-10) NPRS (with 10 as the worse outcome) Area under the curve (AUC)
Time Frame: time 0 to Day 15
Measure: Mean (Standard Deviation); unit: Scores on a scale*hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Scores on a scale*hours
  AUC 0-12 hours | 12.57 (10.26) | 14.25 (7.07) | 29.82 (24.55) | 32.47 (27.95) | 30.07 (31.66) | 41.77 (30.90)
  AUC 12-24 hours | 48.07 (35.69) | 56.70 (30.72) | 78.88 (11.89) | 57.28 (39.58) | 43.98 (23.47) | 79.46 (19.87)
  AUC 24-72 hours | 109.57 (82.15) | 163.48 (108.59) | 169.35 (47.44) | 126.53 (102.53) | 101.62 (63.19) | 215.75 (93.95)
  AUC 24-96 hours | 169.08 (132.37) | 267.47 (177.48) | 251.07 (94.99) | 200.33 (167.29) | 133.70 (84.38) | 348.49 (169.76)
  AUC 24 hours - 1 week | 294.12 (258.23) | 534.62 (423.60) | 512.52 (269.58) | 317.30 (264.28) | 212.07 (144.15) | 718.80 (422.15)
  AUC 24 hours - 2 weeks | 555.60 (583.64) | 1150.53 (1127.42) | 972.87 (816.65) | 561.00 (429.33) | 452.37 (379.82) | 1588.12 (1165.62)

4. Secondary Outcome: Postoperative Use of Analgesics
Description: Use of postoperative analgesic therapy/treatments
  Opioid consumption is recorded on the concomitant medication and/or the rescue medications pages and is calculated as the sum of the morphine milligram equivalents (MEQ) of all the medications recorded as taken during the period. For subjects who discontinued from the efficacy portion of the study, all medications are included regardless of whether they were taken before or after the discontinuation
Time Frame: Daily up through Day 15
Measure: Mean (Standard Deviation); unit: Morphine milligram equivalents (MEQ)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Morphine milligram equivalents (MEQ) | 40.00 (39.02) | 38.17 (39.78) | 68.75 (79.86) | 42.50 (41.53) | 47.50 (47.59) | 94.60 (58.15)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 64 days for participants in the study. This was comprised of a screening period that could be up to 28 days and subsequent clinic visits through Day 29. A Day 36 visit was required only if the wound was not considered healed by Day 29.
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information in this study did not differ from the clinicaltrials.gov definitions.
Groups:
- CA-008 Cohort 1: CA-008 in 0.5 mg
- CA-008 Cohort 2: CA-008 in 1 mg
- CA-008 Cohort 3: CA-008 in 2 mg
- CA-008 Cohort 4: CA-008 in 3 mg
- CA-008 Cohort 5: CA-008 in 4.2 mg
Arm/Group | CA-008 Cohort 1 | CA-008 Cohort 2 | CA-008 Cohort 3 | CA-008 Cohort 4 | CA-008 Cohort 5 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 4/6 | 2/6 | 3/6 | 3/6 | 4/6 | 4/10
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CA-008 Cohort 1 (N=6) | CA-008 Cohort 2 (N=6) | CA-008 Cohort 3 (N=6) | CA-008 Cohort 4 (N=6) | CA-008 Cohort 5 (N=6) | Placebo (N=10)
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT03307837/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT03307837/SAP_001.pdf